CLINICAL TRIAL: NCT02539966
Title: Safety & Performance Study of the FANTOM Sirolimus-Eluting Bioresorbable Coronary Scaffold
Acronym: FANTOM II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: REVA Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCT6200
Record Dates: First submitted 2015-09-01; First posted 2015-09-03 (Estimated); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cohort A (Experimental): Fantom Sirolimus-Eluting Coronary Bioresorbable Scaffold - Treatment Group A (6-month angiographic follow-up)
  Interventions: Device: Fantom Sirolimus-Eluting Coronary Bioresorbable Scaffold
- Cohort B (Experimental): Fantom Sirolimus-Eluting Coronary Bioresorbable Scaffold - Treatment Group B (9-month angiographic follow-up)
  Interventions: Device: Fantom Sirolimus-Eluting Coronary Bioresorbable Scaffold
- Cohort C (Experimental): Fantom Sirolimus-Eluting Coronary Bioresorbable Scaffold - Treatment Group C (6-month angiographic follow-up), Long Lesion/Multi-Vessel
  Interventions: Device: Fantom Sirolimus-Eluting Coronary Bioresorbable Scaffold

INTERVENTIONS:
Device: Fantom Sirolimus-Eluting Coronary Bioresorbable Scaffold — Bioresorbable Drug-Eluting Scaffold Implantation for the Treatment of Coronary Artery Disease

SUMMARY:
The FANTOM II trial is intended to assess safety and performance of the Fantom Bioresorbable Coronary Scaffold in native coronary arteries.

ELIGIBILITY:
Inclusion Criteria:

* Patient has evidence of myocardial ischemia or a positive functional study
* Target lesion has a visually estimated stenosis of ≥50% and <100%
* Target lesion is located in a native coronary artery with average reference vessel diameter ≥ 2.5mm and ≤ 3.5mm
* Lesion length ≤ 20 mm by visual estimate (N/A for Cohort C)
* Baseline TIMI flow ≥ 2

Exclusion Criteria:

* The patient has experienced an acute myocardial infarction (AMI: STEMI or NSTEMI) within 72 hours of the procedure and either CK-MB or Troponin has not returned to within 2X ULN.
* Patient has a left ventricular ejection fraction < 40%
* Patient has unprotected left main coronary disease with ≥50% stenosis
* The target vessel is totally occluded (TIMI Flow 0 or 1)
* Target lesion involves a bifurcation (a lesion with a side branch ≥ 1.5 mm in diameter containing a ≥ 50% stenosis).
* Target lesion is located within a bypass graft
* Target lesion has possible or definite thrombus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2019-08 (Actual); Study Completion 2024-09 (Actual)

PRIMARY OUTCOMES:
Major Adverse Cardiac Events (MACE) - Cohorts A, B and C | 6 months
  Cardiac Death, Myocardial Infarction (Q-Wave, Non Q-wave: CK-MB >5X ULN) (MI), and target lesion revascularization (TLR)
Quantitative Coronary Angiography (QCA) derived parameters - Cohorts A and C | 6 months
  Late Lumen Loss

SECONDARY OUTCOMES:
Quantitative Coronary Angiography (QCA) derived parameters - Cohort B | 9 months
  Late Lumen Loss
Quantitative Coronary Angiography (QCA) derived parameters - Cohorts A and C | 6 months
  Minimum Lumen Diameter (MLD)
Quantitative Coronary Angiography (QCA) derived parameters - Cohort B | 9 months
  Minimum Lumen Diameter (MLD)
Quantitative Coronary Angiography (QCA) derived parameters - Cohorts A and C | 6 months
  % Diameter Stenosis
Quantitative Coronary Angiography (QCA) derived parameters - Cohort B | 9 months
  % Diameter Stenosis
Quantitative Coronary Angiography (QCA) derived parameters - Cohorts A and C | 6 months
  Binary Restenosis
Quantitative Coronary Angiography (QCA) derived parameters - Cohort B | 9 months
  Binary Restenosis
Major Adverse Cardiac Events (MACE) - Cohorts A, B and C | 12, 24, 36, 48 and 60 months
  Cardiac Death, Myocardial Infarction (Q-Wave, Non Q-wave: CK-MB >5X ULN) (MI), and target lesion revascularization (TLR)
Target Lesion Revascularization (TLR) - Cohorts A, B and C | 12, 24, 36, 48 and 60 months
  Percentage of patients with TLR at each time point
Target Vessel Revascularization (TVR) - Cohorts A, B and C | 12, 24, 36, 48 and 60 months
  Percentage of patients with TVR at each time point
Target Vessel Failure (TVF) - Cohorts A, B and C | 12, 24, 36, 48 and 60 months
  Percentage of patients with TVF at each time point
Acute Technical Success - Cohorts A, B and C | Day 0
  Successful acute delivery and deployment of the device
Procedural Success - Cohorts A, B and C | 30 days
  Percentage of patients with angiographic success (final diameter stenosis <50% without occurrence of MACE)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Abizaid, MD, PhD, Principal Investigator — Instituto Dante Pazzanese de Cardiologia; Christoph K Naber, PD Dr. med, Principal Investigator — Elisabeth-Krankenhaus Essen
Locations (28):
- Australia (3):
  - The Prince Charles Hospital, Chermside
  - St Vincent's Hospital Sydney, Darlinghurst
  - Prince of Wales Hospital (Eastern Heart), Randwick
- Cardiovascular Center Aalst, Aalst, Belgium
- Brazil (2):
  - Albert Einstein Hospital, São Paulo
  - Instituto Dante Pazzanese de Cardiologia, São Paulo
- Denmark (3):
  - Aarhus University Hospital (Skejby), Aarhus
  - Rigshospitalet, Copenhagen
  - Odense University Hospital, Odense
- France (4):
  - institut Hospitalier J.Cartier, Massy
  - La Pitié-Salpétrière, Paris
  - Clinique Pasteur, Toulouse
  - Hôpital Rangueil, Toulouse
- Germany (7):
  - Am Urban Hospital, Berlin, Berlin
  - Friedrichshein Hospital, Berlin, Berlin
  - Klinikum Coburg, Coburg
  - St.- Johannes-Hospital Dortmund, Dortmund
  - Universitätsklinikum Erlangen, Erlangen
  - Elisabeth-Krankenhaus Essen, Essen
  - Universitätsklinikum Schleswig-Holstein, Kiel
- Netherlands (4):
  - Academic Medical Center Amsterdam, Amsterdam
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Erasmus Medical Center, Rotterdam
  - University Medical Center Utrecht, Utrecht
- Poland (4):
  - Krakowskie Centrum Kardiologii Inwazyjnej, Krakow
  - Szpital Uniwersytecki w Krakowie, Krakow
  - Szpital Kliniczny Przemienienia Panskiego UM w Poznaniu, Poznan
  - Oddział Kardiologii Inwazyjnej I Katedra, Warsaw

REFERENCES:
- [Derived] Chevalier B, Abizaid A, Carrie D, Frey N, Lutz M, Weber-Albers J, Dudek D, Weng SC, Akodad M, Anderson J, Stone GW. Clinical and Angiographic Outcomes With a Novel Radiopaque Sirolimus-Eluting Bioresorbable Vascular Scaffold. Circ Cardiovasc Interv. 2019 Jun;12(6):e007283. doi: 10.1161/CIRCINTERVENTIONS.118.007283. Epub 2019 Jun 10. PMID 31177821